CLINICAL TRIAL: NCT06551012
Title: The Influence of Active Muscle Mass and Nitrate Supplementation on Fatigability in Individuals With Heart Failure
Brief Title: Neuromuscular Fatigability in Individuals With Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Principal Investigator, Callum Brownstein, Lecturer in Exercise Physiology, Newcastle University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 340538
Record Dates: First submitted 2024-07-25; First posted 2024-08-13 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Exercise; Physiology; Fatigability
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomised, cross-over trial. Participants will perform exercise following consumption of nitrate-rich beetroot juice and beetroot juice with nitrate extracted
Who Masked: Participant, Investigator
Masking Description: The study will be double-blinded, with participant and investigator unaware of the treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate-rich beetroot juice (Experimental): Participants will consume 2 x 70 ml bottles of nitrate-rich beetroot juice for a 7 day period prior to exercise testing
  Interventions: Dietary Supplement: Nitrate-rich beetroot juice
- Beetroot juice with nitrate extracted (Placebo Comparator): Participants will consume 2 x 70 ml bottles of beetroot juice with nitrate extracted for a 7 day period prior to exercise testing
  Interventions: Dietary Supplement: Beetroot juice with nitrate extracted

INTERVENTIONS:
Dietary Supplement: Nitrate-rich beetroot juice — Participants will consume 2 x 70 ml bottles of nitrate-rich beetroot juice for a 7 day period prior to exercise testing
  Arms: Nitrate-rich beetroot juice
Dietary Supplement: Beetroot juice with nitrate extracted — Participants will consume 2 x 70 ml bottles of beetroot juice with nitrate extracted for a 7 day period prior to exercise testing
  Arms: Beetroot juice with nitrate extracted

SUMMARY:
Brief summary

The aims of this project are to 1) characterise muscle fatigue in individuals with chronic heart failure during exercise involving a smaller and larger muscle mass (Part I), 2) to determine the effect of nitrate supplementation on muscle fatigue during large muscle mass exercise in individuals with chronic heart failure (Part II), 3) understand the impact of exercise intolerance on quality of life in individuals with chronic heart failure (Part III). The main questions it aims to answer are:

* Is muscle fatigue attenuated during exercise engaging a smaller vs larger muscle mass in individuals with chronic heart failure owing to lower central cardiopulmonary constraints?
* Can supplementation with nitrate-rich beetroot juice reduce muscle fatigue and/or accelerate post-exercise recovery of muscle function in response to whole body exercise in individuals with heart failure?
* What impact does exercise intolerance have on the lives of individuals with chronic heart failure?

For Part I, researchers will compare muscle fatigue during single- and double-leg incremental cycling in individuals with chronic heart failure.

For Part II, researchers will compare muscle fatigue in individuals with chronic heart failure during double-leg incremental cycling following a period of beetroot juice supplementation containing nitrate, or with a placebo drink consisting of beetroot juice with nitrate extracted.

For Part III, semi-structured interviews will be conducted to investigate the symptoms associated with performing physical activity and on the impact of exercise intolerance on quality of life in individuals with chronic heart failure.

DETAILED DESCRIPTION:
Background:

Exercise intolerance is a hallmark symptom of chronic heart failure with reduced ejection fraction (HFrEF) and is associated with reduced quality of life as well as being a strong prognostic indicator. Research in recent years has attempted to better understand the aetiology of exercise intolerance to provide therapeutic targets to improve physical capacity and quality of life, with studies primarily focusing on maximal oxygen uptake, metabolic thresholds and oxygen uptake kinetics. Another important determinant of exercise intolerance is neuromuscular fatigability, defined as the reduction in neuromuscular function measured after exercise of a discrete time period. At present, the few studies that have assessed neuromuscular fatigability in individuals with HFrEF have utilised exercise involving a small muscle mass, such as isometric knee extension. However, one limitation of this approach is that it does not reflect the types of activity performed on a daily basis, and thereby lacks ecological validity. Specifically, activities of daily living (e.g. walking, gardening, housework or climbing stairs) involve dynamic, large muscle mass exercise and in turn a substantially higher cardiorespiratory demand relative to isometric tasks. At present, there is limited research assessing neuromuscular fatigability in individuals with HFrEF during large muscle mass exercise. Research characterising fatigability and determining its underlying mechanisms can help better understand the aetiology of exercise intolerance, and in turn provide therapeutic targets aimed at improving physical capacity and quality of life in individuals with HFrEF.

Neuromuscular fatigability is tightly linked with oxygen transport, with impairments in oxygen transport associated with a higher reliance on anaerobic metabolism and the production of contractile function-impairing metabolites. Given that HFrEF is associated with impairments at multiple steps along the oxygen cascade, limitations in oxygen transport likely represent an important contributor to neuromuscular fatigability in individuals with HFrEF. In turn, the loci of limitations in oxygen transport can be broadly categorised as being of central (cardiac and/or pulmonary) and peripheral origin (vascular and muscle mitochondrial). While those with HFrEF may exhibit higher neuromuscular fatigability as a result of both central and peripheral impairments, the relative importance of each is uncertain. An experimental model which has previously been used to provide insight into central and peripheral determinants of neuromuscular fatigability is through the manipulation of active muscle mass during exercise. Performing exercise with a smaller muscle mass, such as during single-leg cycling (SLC), allows a cardiac and pulmonary reserve to become available, meaning that cardiac and pulmonary constraints to exercise tolerance are attenuated. The lower cardiopulmonary constrains on leg blood flow and oxygen delivery in SLC will therefore permit the assessment of neuromuscular fatigability with a lower influence of central limitations. In contrast, when exercising with a large muscle mass, such as during double-leg cycling (DLC), there is a greater oxygen demand as a larger proportion of the total bodily muscle mass is active. As such, the contribution of impaired cardiac output in individuals with HFrEF becomes of greater relative importance during large muscle mass exercise. Moreover, the increased demand of respiration during large muscle mass exercise requires greater redistribution of blood and oxygen centrally, away from the exercising muscles. Comparing responses to SLC and DLC can therefore provide insight into the relative contribution of central and peripheral limitations to neuromuscular fatigue and exercise intolerance in those with HFrEF.

One potential strategy to attenuate fatigability is through nitrate supplementation (i.e. beetroot juice). Specifically, the consumption of nitrate-rich beetroot juice promotes increased nitric oxide bioavailability, which in turn can enhance local perfusion and oxygenation, skeletal muscle contractility, and muscle efficiency. Given that individuals with CHF have impaired nitric oxide bioavailability and reduced local perfusion and oxygenation, which likely contribute to impaired fatigability, nitric oxide represents an attractive intervention to mitigate fatigability and improve exercise tolerance. To date, no study has assessed the effect of nitrate supplementation on neuromuscular fatigability in individuals with CHF.

Aims:

The aims of this project are to 1) characterise muscle fatigue in individuals with chronic heart failure during exercise involving a smaller and larger muscle mass (Part I), 2) to determine the effect of nitrate supplementation on muscle fatigue during large muscle mass exercise in individuals with chronic heart failure (Part II), 3) understand the impact of exercise intolerance on quality of life in individuals with chronic heart failure (Part III).

Study design:

Part I is a cross-sectional, observational study, which will characterise neuromuscular fatigability in individuals with HFrEF during DLC and SLC. On seperate visits and in a randomised order, participants will perform incremental SLC and DLC to exhaustion, with cycling interspersed with measures of neuromuscular function. Part II is a randomised crossover interventional study, which will assess neuromuscular fatigability following nitrate supplementation and a placebo-control in individuals with HFrEF during DLC. For part II, participants will consume nitrate-rich beetroot juice in the lead up to one visit, and beetroot juice with nitrate extracted as a placebo-control in the lead up to another visit, with the order of the conditions randomised. Part III is a qualitative study, which will evaluate the impact of exercise intolerance on quality of life in individuals with HFrEF through semi-structured interviews and questionnaires. All participants will complete both Parts I and II of the study, while Part III is optional (i.e. participants will be able to participate in Parts II and II if they choose not to take part in Part III).

Recruitment procedures:

Patients will be identified from the Heart Failure Clinic run at the Royal Victoria Infirmary and Freeman Hospital, Newcastle upon Tyne, by Consultant Cardiologists. The consultant cardiologist will then invite the patient to talk to a member of the research team. This will take place at the end of the patient's consultation, after which a member of the research team will meet the patient to explain the study. If the patient is interested, they will be provided with an information sheet. To avoid coercion, the patient will not be asked to make a decision in the presence of a member of the research team, and instead will be afforded 48 hours to read the information sheet and decide whether they would like to participate. The research team will request to call the patient after this 48 hour period to discuss the study and answer any questions. If the patient is happy to proceed when they will be invited to the Clinical Research Facility for Visit 1, where they will provide informed consent if they are willing to become a participant in the study.

Research visits - Parts I and II - Quantitative work package:

Individuals with HFrEF (n = 28) will visit the NIHR Clinical Research Facility on 4 occasions across Parts I and II of the study. Visit 1 will involve screening and consent, completion of questionnaires, familiarisation with study procedures, and performing a non-invasive measurement of mitochondrial function using near-infrared spectroscopy (NIRS). Visits 2-4 will be randomised in order, and will include, 1) incremental single-leg cycling to exhaustion with intermittent assessments of neuromuscular function, 2) incremental double-leg cycling to exhaustion with intermittent assessments of neuromuscular function, following a period of supplementation with nitrate-rich beetroot juice and, 3) incremental double-leg cycling to exhaustion with intermittent assessments of neuromuscular function, following a period of supplementation with a nitrate-extracted beetroot juice placebo.

Part III - Qualitative work package:

While Parts I and II will further our understanding on the aetiology of exercise intolerance and the effect of nitrate supplementation in improving exercise tolerance in individuals with CHF, it is important to clarify the impact of exercise intolerance on the lives of these individuals. As such, the aim of Part III is to understand the symptoms associated with performing exercise and the impact of exercise intolerance on social, functional and emotional functioning on individuals with CHF.

One optional semi-structured interviews will be conducted with the participants who provide consent to participate in this part of the study (n = 28 or until saturation in findings) once they have completed the Parts I and II. Participants may choose to opt out from this part of the study and this option will be included in the consent form. An interview specific topic guide has been developed on symptoms associated with performing physical activity and on the impact of exercise intolerance on quality of life. Data from the semi-structured interviews will be analysed thematically using an inductive approach. All interviews will be transcribed verbatim. The interviews will be conducted remotely and participants will be given the option to use the zoom platform or receive a telephone call.

Sample size and statistical analysis:

The target sample size is based on a power calculation using the expected effect moderate effect size for a positive effect of nitrate supplementation on exercise tolerance derived from previous research. For an a of 0.05 and a power of 0.80, a total sample size of 24 is required. To account for potential drop-outs, an additional 4 participants will be recruited, based on drop-out rate of ~20% in studies assessing the effect of nitrate supplementation on exercise tolerance. For Part I, the analysis will include a two-way repeated measures analysis of variance (ANOVA) to determine the effect of the magnitude of active muscle mass (small vs. large) on neuromuscular fatigability and other physiological variables measured during cycling. For Part II, the analysis will include a two-way repeated measures ANOVA to determine the effect of nitrate supplementation vs. placebo on neuromuscular fatigability and other physiological variables measured during cycling. For Part III, an inductive approach to analysis will be made and data saturation of themes will be determined at the analysis stage. Two independent reviewers in the research study team will code and extract segments of the data to identify key themes. Inclusion of supporting quotes from each of the themes will be included in the write up and publication.

Funding:

The study is funded through a studentship offered by the Faculty of Medical Sciences, Newcastle University.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a left ventricular ejection fraction < 40% who have been diagnosed for at least 3 months.
* Classified according to New York Heart Association (NYHA) class II-III.
* Clinically stable and receiving optimal medical treatment.
* Aged ≥ 45 years old.
* Ability to read, write and converse in English without the support of an interpreter.
* Willingness to undertake physical activity with no contraindications to physical activity and capable of performing activities of daily living independently, without the use of a walking aid.
* Able to provide written informed consent.

Exclusion Criteria:

* An electrically implanted device (e.g., pacemaker, left ventricular assist device).
* Uncontrolled cardiac arrhythmias, myocardial infarction, percutaneous coronary intervention and/or bypass graft surgery up to 3 months previously.
* Receiving antacids or proton pump, xanthine oxidase, or phosphodiesterase inhibitors which affect the reduction of nitrate to nitrite and nitrite to nitric oxide.
* Treated with organic nitrates (e.g., trinitroglycerin)
* Major multi-morbidity or other alternative diagnoses of no obvious acute and self-limiting cause (e.g., patients with a terminal diagnosis of cancer, patients in receipt of oxygen therapy or oxygen saturation at rest <92%).
* Obesity (body mass index > 30 kg/m2).
* Current smoker.
* Presented with severe symptoms requiring urgent assessment and stabilisation (e.g., breathlessness at rest, hypotension, confusion).
* Severe physical disability preventing them from functioning independently;
* Unable to provide informed consent.
* Currently taking part in any other study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Maximal voluntary contraction force | 3 years
  Maximal voluntary contraction (MVC) force of the right knee extensor will be taken pre, during and post-exercise.

SECONDARY OUTCOMES:
Voluntary activation | 3 years
  Voluntary activation (%) will be measured using supramaximal femoral nerve stimulation during maximal voluntary contractions at pre, during and post-exercise.
Resting evoked twitch force | 3 years
  Resting evoked twitch force (Newtons) will be measured using supramaximal femoral nerve stimulation following maximal voluntary contractions at pre, during and post-exercise.
Electromyography | 3 years
  Electromyography (root mean squared) of vastus lateralis measured throughout exercise
Time constant for recovery of muscle oxygen uptake | 3 years
  Non-invasive measure of skeletal muscle oxidative capacity measured using NIRS-derived time constant for recovery of muscle oxygen uptake
Microvascular responsiveness | 3 years
  A 5 minute period of occlusion will be used, followed by deocclusion. Using NIRS, the slope of the increase in oxygenated haemoglobin following deocclusion by will quantified through the upslope of a 10 s window following cuff release.
Cardiac output | 3 years
  Cardiac output (L/min) will be assessed throughout exercise using Bioreactance technology
Stroke volume | 3 years
  Stroke volume (ml/min) will be assessed throughout exercise using Bioreactance technology
Heart rate | 3 years
  Heart rate (bpm) will be assessed throughout exercise using Bioreactance technology
Mean arterial blood pressure | 3 years
  Mean arterial blood pressure (mmHg) will be assessed throughout exercise using Bioreactance technology
Oxygen consumption | 3 years
  Oxygen consumption (ml/kg/min) will be measured throughout exercise using a metabolic analyser
Carbon dioxide production | 3 years
  Carbon dioxide production (ml/min) will be measured throughout exercise using a metabolic analyser throughout exercise
Ventilation | 3 years
  Ventilation (L/min) will be measured throughout exercise using a metabolic analyser throughout exercise
Carbon dioxide ventilatory equivalent | 3 years
  Litres of ventilation per litre of carbon dioxide production (Ve/VCO2) will be measured throughout exercise using a metabolic analyser throughout exercise
Tissue oxygen saturation | 3 years
  Measurements of tissue oxygen saturation (%) taken from near-infrared spectroscopy throughout exercise
Deoxygenated haemoglobin | 3 years
  Measurements of deoxygenated haemoglobin (%) will be taken from near-infrared spectroscopy throughout exercise

CONTACTS AND LOCATIONS:
Overall Officials: Callum Brownstein, PhD, Principal Investigator — Newcastle University

IPD SHARING:
Plan to Share IPD: Yes
Data archive and sharing Research data that supports publications and unpublished data of value at project end will be archived with supporting documentation in data.ncl (https://data.ncl.ac.uk/), Newcastle's Research Data Repository. The datasets will be made public under a Creative Commons licence to ensure credit is given when the data is reused and access provided for at least ten years. Data deposited will also be assigned a persistent identifier (i.e. DOI) that can be included in project outputs, including publications, to detail how and where the data can be accessed. At this stage all study identification numbers will be removed and all data will be anonymised before being archived and shared through the repository. Where there is a risk to data being re-identified the dataset will be archived to make the record findable but access will be controlled and dependent on the future use of the data in question.
Time Frame: 5 years
URL: https://data.ncl.ac.uk/

REFERENCES:
- [Background] Swank AM, Horton J, Fleg JL, Fonarow GC, Keteyian S, Goldberg L, Wolfel G, Handberg EM, Bensimhon D, Illiou MC, Vest M, Ewald G, Blackburn G, Leifer E, Cooper L, Kraus WE; HF-ACTION Investigators. Modest increase in peak VO2 is related to better clinical outcomes in chronic heart failure patients: results from heart failure and a controlled trial to investigate outcomes of exercise training. Circ Heart Fail. 2012 Sep 1;5(5):579-85. doi: 10.1161/CIRCHEARTFAILURE.111.965186. Epub 2012 Jul 6. PMID 22773109
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Poole DC, Hirai DM, Copp SW, Musch TI. Muscle oxygen transport and utilization in heart failure: implications for exercise (in)tolerance. Am J Physiol Heart Circ Physiol. 2012 Mar 1;302(5):H1050-63. doi: 10.1152/ajpheart.00943.2011. Epub 2011 Nov 18. PMID 22101528
- [Background] Hepple RT. The role of O2 supply in muscle fatigue. Can J Appl Physiol. 2002 Feb;27(1):56-69. doi: 10.1139/h02-004. PMID 11880691
- [Background] Weavil JC, Thurston TS, Hureau TJ, Gifford JR, Kithas PA, Broxterman RM, Bledsoe AD, Nativi JN, Richardson RS, Amann M. Heart failure with preserved ejection fraction diminishes peripheral hemodynamics and accelerates exercise-induced neuromuscular fatigue. Am J Physiol Heart Circ Physiol. 2021 Jan 1;320(1):H338-H351. doi: 10.1152/ajpheart.00266.2020. Epub 2020 Nov 8. PMID 33164549
- [Background] Jones TW, Houghton D, Cassidy S, MacGowan GA, Trenell MI, Jakovljevic DG. Bioreactance is a reliable method for estimating cardiac output at rest and during exercise. Br J Anaesth. 2015 Sep;115(3):386-91. doi: 10.1093/bja/aeu560. Epub 2015 Feb 6. PMID 25659999
- [Background] Jones AM, Ferguson SK, Bailey SJ, Vanhatalo A, Poole DC. Fiber Type-Specific Effects of Dietary Nitrate. Exerc Sport Sci Rev. 2016 Apr;44(2):53-60. doi: 10.1249/JES.0000000000000074. PMID 26829247
- [Background] Coggan AR, Broadstreet SR, Mahmood K, Mikhalkova D, Madigan M, Bole I, Park S, Leibowitz JL, Kadkhodayan A, Thomas DP, Thies D, Peterson LR. Dietary Nitrate Increases VO2peak and Performance but Does Not Alter Ventilation or Efficiency in Patients With Heart Failure With Reduced Ejection Fraction. J Card Fail. 2018 Feb;24(2):65-73. doi: 10.1016/j.cardfail.2017.09.004. Epub 2017 Sep 12. PMID 28916479

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT06551012/Prot_SAP_000.pdf